CLINICAL TRIAL: NCT00019929
Title: Phase II Trial of Individualized Mutant p53 Peptide-Pulsed Cultured Autologous Dendritic Cells in the Adjuvant Treatment of Patients With Locally Advanced Non-Small Cell Lung Cancer After Standard Therapy
Brief Title: Vaccine Therapy in Treating Patients With Stage III Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067284; NCI-99-C-0142; VU-VCC-THO-9814; NCI-T96-0045; NCT00001829 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2005-11

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Chemotherapy, Adjuvant

INTERVENTIONS:
Biological: mutant p53 peptide pulsed dendritic cell vaccine
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: This phase II trial is studying vaccine therapy given after standard therapy to see how well it works in treating patients with stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the overall survival in patients with locally advanced non-small cell lung cancer immunized with adjuvant mutant p53 peptide-pulsed autologous dendritic cells after standard therapy.
* Assess the safety and immunological efficacy of this regimen in terms of inducing or boosting a mutant p53-specific immune response in this patient population.

OUTLINE: Patients undergo p53 gene mutation analysis. Patients without a suitable gene mutation receive no vaccination. Patients with a suitable p53 gene mutation receive mutant p53 peptide-pulsed autologous dendritic cells IV over 1-2 minutes weekly for 5 weeks. Patients achieving an immune response with no evidence of progressive disease may receive additional vaccinations every 2 months for a maximum of 10 immunizations.

Patients are followed for 5 years.

PROJECTED ACCRUAL: Approximately 120 patients (40 on the vaccination arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IIIA or IIIB non-small cell lung cancer (NSCLC) with one of the following p53 mutations:

  * Point mutation altering the protein sequence
  * Frame-shift mutation with the generation of a novel sequence
* No significant pleural effusions visible on plain chest radiography
* Must have completed or plan to undergo curative intent therapy for NSCLC

  * At least 2 courses of neoadjuvant chemotherapy for patients with known N2 or N3 resectable disease OR
  * At least 55 Gy radiotherapy with concurrent or sequential chemotherapy for patients with unresectable disease
  * Patients with incidental N2 or N3 disease at time of surgery may receive optional adjuvant chemotherapy and radiotherapy

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Lymphocyte count greater than 475/mm^3
* Granulocyte count greater than 1,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 2.0 mg/dL
* SGOT less than 3 times normal
* Albumin at least 3.0 g/dL
* No signs of acute hepatitis B infection

  * Hepatitis B surface antigen positive allowed provided there are no signs of chronic active hepatitis
* No prior hepatitis C infection

Renal:

* Creatinine less than 2.5 mg/dL
* Calcium less than 11.0 mg/dL (corrected for albumin)

Cardiovascular:

* No myocardial infarction or significant ventricular arrhythmias within the past 6 months

Other:

* No other malignancy within the past 5 years unless curatively treated and probability of recurrence is less than 5%
* HIV negative
* No psychiatric or other condition that would preclude study
* No serious ongoing infection
* No other serious medical condition that would limit life expectancy to less than 2 years
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy and no anticipated need for chemotherapy for at least 2 months after vaccinations

Endocrine therapy:

* At least 4 weeks since prior supraphysiologic steroids and no anticipated need for steroid therapy for at least 2 months after vaccinations

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and no anticipated need for radiotherapy for at least 2 months after vaccinations

Surgery:

* See Disease Characteristics

Other:

* No influenza vaccination if egg allergy present
* At least 4 weeks and no greater than 24 weeks since completion of all prior modalities for primary therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-08; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Disease-free survival by CTEP CTC v2.x
Overall survival by CTEP CTC v2.x
Toxicity by CTEP CTC v2.x

SECONDARY OUTCOMES:
Immunological response by ELISPOT before and 2 weeks after last vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Jay A. Berzofsky, MD, PhD, Study Chair — NCI - Vaccine Branch
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Background] Read EJ, Carter CS, Lee J, et al.: Clinical scale preparation of antigen-pulsed mature autologous dendritic cells for tumor-specific immunotherapy. [Abstract] ISHAGE 2001 Seventh Annual Symposium A-100, 2001.